CLINICAL TRIAL: NCT06553040
Title: The Effect of Albumin Value, HALP Score, and LCR Value on Predicting Survival and Recurrence in Patients With Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Tufan Gumus, Specialist, Ege University
Other Study IDs: EUTFHALPSCOREFORPANCREAS
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Neoplasms; Pancreas Cancer
Keywords: Pancreatic adenocancer; albumin; hemoglobin; lymphocyte; platelet
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate whether the albumin value and the ratios of biochemical markers; hemoglobin, albumin, lymphocyte and platelet (HALP score) and lymphocyte-C-reactive protein ratio (LCR) can predict the survival and recurrence of the disease in patients with pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Whipple operation and total pancreatectomy due to pathologically confirmed pancreatic adenocarcinoma

Exclusion Criteria:

* Patients with other malignant tumors (choledochal tumor, papilla tumor and duodenal tumor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 87 patients who underwent either pancreaticoduodenectomy (Whipple or total pancreatectomy) operations for pancreatic adenocarcinoma in the General Surgery Clinic of Ege University Hospital between January 2017 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival Times | 4 Years
HALP Score | 4 Years
  Hemoglobin x Albumin x Lymphocyte / Platelet
Overall Survival Time | 4 Years
LCR Score | 4 Years
  Lymphocyte / CRP